CLINICAL TRIAL: NCT05392452
Title: Fully Closed-Loop Insulin Delivery in Abdominal Surgery: a Randomised Controlled Two-centre Trial (CLAB-Study)
Brief Title: Fully Closed-Loop Insulin Delivery in Abdominal Surgery (CLAB)
Acronym: CLAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lia Bally (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Lia Bally, Head of Nutrition, Metabolism and Obesity and Head of Research, Insel Gruppe AG, University Hospital Bern
Organization: Insel Gruppe AG, University Hospital Bern (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAB
Record Dates: First submitted 2022-03-25; First posted 2022-05-26 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Perioperative Hyperglycaemia; Insulin Therapy; Elective Surgery; Closed-Loop Glucose Control; Artificial Pancreas; Liver Diseases; Diabetes Mellitus, Type 2; Colon Disease; Gastric Disease; Pancreatic Disease
Keywords: Perioperative Hyperglycaemia; Insulin Therapy; Elective Surgery; Closed-Loop Glucose Control; Artificial Pancreas; Liver Diseases; Diabetes Mellitus, Type 2; Colon Disease; Gastric Disease; Pancreatic Disease
MeSH Terms: conditions — Liver Diseases; Diabetes Mellitus, Type 2; Colonic Diseases; Stomach Diseases; Pancreatic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed-loop insulin therapy (Experimental): Intervention:
  Use of a fully-automated closed-loop insulin delivery system from day of admission until hospital discharge (or maximum 20 days).
  Interventions: Device: CamAPS HX
- Standard insulin therapy (Active Comparator): The control group will receive insulin therapy in accordance with local practice. The insulin regimen during the study period may involve subcutaneous and/or insulin intravenous insulin administration. The modality of insulin treatment, dose adjustment and frequency of glucose monitoring will be at the discretion of the clinical team. No active treatment optimisation will be undertaken by the study team. Participants in the control group will be fitted with the identical study CGM system. The CGM system will be blinded upon hospital admission.
  Interventions: Drug: Standard insulin therapy

INTERVENTIONS:
Device: CamAPS HX — Fully automated closed-loop subcutaneous insulin delivery system. A model predictive controller modulates insulin delivery every 10-12 minutes based on interstitial glucose measurements.
  Arms: Closed-loop insulin therapy
Drug: Standard insulin therapy — Standard insulin therapy according to local clinical practice.
  Arms: Standard insulin therapy

SUMMARY:
The purpose of the study is to assess the efficacy, safety and usability of perioperative fully-automated closed-loop insulin delivery versus standard insulin therapy in patients with diabetes other than type 1 diabetes undergoing elective major abdominal surgery.

DETAILED DESCRIPTION:
The prevalence of diabetes and hyperglycaemia in surgical patients is rising and associated not only with greater complication rates, length of stay, morbidity and mortality rates, but also increased hospital costs and readmission rates. Due to the complex interaction of organs involved in glucose homeostasis (e.g. liver, pancreas) and the frequent need for nutrition support, patients undergoing major abdominal surgery are particularly prone to develop dysglycaemia. While there are guidelines for perioperative glucose management, implementation is challenging and inconsistent. Main reasons are lack of resources, clinical inertia based on fear of hypoglycaemia and multiple handovers between teams.

Closed-loop glucose control represents an emerging diabetes treatment modality that autonomously adjusts insulin delivery according to continuously measured glucose levels. The use of fully automated closed-loop insulin delivery may represent an easy-to-adopt approach for safe and effective perioperative diabetes management. In previous work, the investigators demonstrated that fully closed-loop insulin delivery in adults with type 2 diabetes undergoing various elective surgeries (abdominal, vascular, neurologic, orthopaedic, thoracic) improved glycaemic control by increasing time spent in the glycaemic target range, lowering mean sensor glucose and glycaemic variability without increasing the risk of hypoglycaemia.

In this follow-up trial the investigators will focus on patients undergoing major elective abdominal surgery to further explore the potential of the fully automated closed-loop approach to accommodate the complex needs of this population. Involvement of a second study centre and hospital staff for device management will further allow to assess the usability of the fully closed-loop system for larger multi-centre clinical trials as well as readiness to use the approach in usual clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or over
* Pre-existing or anticipated (surgery-induced) diabetes other than type 1 diabetes
* Expected to require insulin treatment in the perioperative period
* Planned for elective major abdominal surgery at the University Hospital Bern or Basel expected to last ≥ 90 minutes, defined as colorectal, pancreatic, gastric (except bariatric surgery) and hepatic (≥ 2 segments) surgery

Exclusion Criteria:

* Physical or psychological condition likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
* Likely discharge earlier than 72 hours
* Known or suspected allergy to insulin used in this clinical trial
* Type 1 diabetes
* Pregnancy, planned pregnancy, or breast feeding
* Lack of safe contraception for female participants of childbearing potential for the entire study duration (medically reliable method of contraception are considered oral, injectable, or implantable contraceptives, intrauterine contraceptive devices, or any other methods judged as sufficiently reliable by the investigator in individual cases).
* Medically documented allergy towards the adhesive (glue) of plasters or unable tolerate tape adhesive in the area of sensor placement
* Serious skin diseases located at places of the body, which potentially are possible to be used for localisation of the glucose sensor
* Illicit drug abuse or prescription drug abuse
* Incapacity to give informed consent
* Not willingness to wear study devices 24/7
* Not literate in German

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
The proportion of time spent in the target glucose range from 5.6 to 10.0 mmol/L | Assessed from hospital admission until a maximum of 20 days following surgery
  The outcome is based on sensor glucose levels

SECONDARY OUTCOMES:
Proportion of time spent with sensor glucose values above target (> 10.0 mmol/L) | Assessed from hospital admission until a maximum of 20 days following surgery
  The outcome is based on sensor glucose levels
Proportion of time spent with sensor glucose <3.0 mmol/L | Assessed from hospital admission until a maximum of 20 days following surgery
  The outcome is based on sensor glucose levels
Proportion of time spent with sensor glucose < 3.9 mmol/L | Assessed from hospital admission until a maximum of 20 days following surgery
  The outcome is based on sensor glucose levels
Average of sensor glucose level | Assessed from hospital admission or until a maximum of 20 days following surgery
  The outcome is based on sensor glucose levels
Proportion of time spent with sensor glucose below target (< 5.6 mmol/L) | Assessed from hospital admission until a maximum of 20 days following surgery
  The outcome is based on sensor glucose levels
Standard deviation of sensor glucose levels | Assessed from hospital admission or until a maximum of 20 days following surgery
  The outcome is based on sensor glucose levels
Coefficient of variation of sensor glucose levels | Assessed from hospital admission until a maximum of 20 days following surgery
  The outcome is based on sensor glucose levels
Total daily insulin dose | Assessed from hospital admission until a maximum of 20 days following surgery
  Insulin dose received by the patients in units/24h
Post-surgery comorbidity | Assessed at 30 days following surgery
  Assessed using the Comprehensive Complication Index (CCI)
Length of hospital stay | Up to 20 days
  Assessed based on the information in electronic health records
Peri- and postoperative costs (perspectives: hospital, statutory health insurance system) | Assessed from hospital admission until a maximum of 30 days following surgery
  Assessed based on the information from device manufacturers, hospital administration system and standard external sources for healthcare utilisation unit costs.

OTHER OUTCOMES:
Number of severe hypoglycaemia (< 2.2 mmol/L) | Assessed from hospital admission until a maximum of 20 days following surgery
  Based on point-of-care capillary measurements. This is a safety outcome.
Number of clinically significant hyperglycaemic events (>20.0 mmol/L) with ketonaemia (beta-hydroxybutyrate >1.0 mmol/L) | Assessed from hospital admission until a maximum of 20 days following surgery
  Based on point-of-care capillary measurements. This is a safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: Lia Bally, MD PhD, Principal Investigator — Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Inselspital, Bern University, Unviersity of Bern; Thierry Girard, MD, Principal Investigator — Anaesthesiology, University Hospital Basel
Locations (2):
- Switzerland (2):
  - Anaesthesiology, University Hospital Basel, Basel
  - Department of Diabetes, Endocrinology, Clinical Nutrition and Metabolism, Inselspital, Bern University Hospital, Bern